CLINICAL TRIAL: NCT06899568
Title: Finite Element Evaluation of Patient Specific Z-shaped Plate With Lingual Extension Versus Conventional Two Mini Plates for Mandibular Parasymphyseal Fracture Fixation
Brief Title: Finite Element and z Shap Mini Plate With Lingual Extension
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohsen, associate professor, Fayoum University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3333
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Mandible Fracture
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- z miniplate with lingual extension (Experimental)
  Interventions: Procedure: z mini plate with lingual extension
- two mini plate (Active Comparator)
  Interventions: Procedure: two mini plates

INTERVENTIONS:
Procedure: z mini plate with lingual extension — parasympheseal fracture model fixed with z mini plate with lingual extension
  Arms: z miniplate with lingual extension
Procedure: two mini plates — parasympheseal fracture model fixed with conventional 2 mini plates
  Arms: two mini plate

SUMMARY:
* A cone beam CT (CBCT) scan of the patient, will be used to create a 3D scanned image of parasympheseal mandibular fracture
* 3D images will be introduced to finite element (FA)software to evaluate Stresses (MPa) and Life time (cycle) For each model and determine which plate is the best

ELIGIBILITY:
Inclusion Criteria:

- parasymhyseal fracture

Exclusion Criteria:

• absence of other facial trauma, mandibular condylar fracture

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2025-04-27 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-27 (Estimated)

PRIMARY OUTCOMES:
stress on the plate will be measured for each point of application by finite element (FA) software | immediate after the procedure

IPD SHARING:
Plan to Share IPD: Undecided